CLINICAL TRIAL: NCT06427252
Title: The Efficacy and Safety of HIPEC Combined With PD-1 and SOX Chemotherapy for the Translational Treatment of Gastric or Esophagogastric Junctional Cancer With Peritoneal Metastasis: A Prospective, Multicenter Phase II Study
Brief Title: The Efficacy and Safety of HIPEC Combined With PD-1 and SOX Chemotherapy for the Translational Treatment of GC or EGJC With PM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HISTORIA
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer, Metastatic
Keywords: gastric cancer; peritoneal metastasis; HIPEC; immunotherapy
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HIPEC plus PD-1 plus SOX therapy (Experimental): HIPEC treatment (paclitaxel, at 43°C for 60 min) was performed on the 1st day after the first exploratory laparotomy and on the third day after the radical surgery for a total of 2-3 times (total amount of paclitaxel was 175 mg/m2 ). Systemic therapy was started 3 weeks after HIPEC. Systemic therapy including: Tirilizumab: 200 mg, Q3W; oxaliplatin: 130mg/m2, Q3W; Herceptin: loading dose of 8 mg/kg followed by 6 mg/kg Q3W. Tegeo: Oral administration: 40 mg per dose for BSA <1.25, 50 mg per dose for BSA 1.25 to 1.5, and 60 mg per dose for BSA ≥1.5, twice daily for each treatment cycle Q3W; After 2-6 weeks, laparoscopic exploration was performed, PCI score was calculated, and radical surgery was performed in patients who were eligible for radical surgery. Postoperative HIPEC was performed twice.
  Interventions: Drug: HIPEC; Drug: Systemic therapy

INTERVENTIONS:
Drug: HIPEC — In the experimental group, HIPEC treatment (paclitaxel, 3000 ml of physiological saline at 43°C for 60 min) was performed on the first day after the first exploratory laparotomy and on the third day after the radical surgery for a total of 2-3 times (total amount of paclitaxel was 175 mg/m2 ), with an interval of not more than 72 h. Intravenous systemic therapy was started 3 weeks after the completion of HIPEC treatment. systemic therapy.
Drug: Systemic therapy — 1. Tirilizumab: 200 mg, i.v., D1, Q3W;
  2. oxaliplatin: 130mg/m2, i.v., D1, Q3W;
  3. Herceptin: a tri-weekly dosing regimen with an initial loading dose of 8 mg/kg followed by 6 mg/kg Q3W.
  4. Tegeo: Oral administration: 40 mg per dose for BSA <1.25, 50 mg per dose for BSA 1.25 to 1.5, and 60 mg per dose for BSA ≥1.5, twice daily for each treatment cycle D1-D14, Q3W;

SUMMARY:
Gastric cancer (GC) with peritoneal metastasis has a poor prognosis and short survival. In recent years, heat intraperitoneal perfusion chemotherapy (HIPEC) has gained better efficacy in the treatment of peritoneal metastases of many malignant tumors, including GC with peritoneal metastasis. The use of immune checkpoint inhibitors (ICIs) in the treatment of advanced GC has made significant progress in recent years. And studies showed that patients who were responded to immunotherapy combined with chemotherapy as the first-line treatment were able to achieve significant survival benefit after radical resection. However, whether HIPEC combined with immunotherapy for peritoneal metastatic gastric cancer improves the R0 resection rate and prolongs survival time is currently unclear. Therefore, we conducted this prospective multicenter clinical trial to explore the effective dose and safety of the combination of systemic chemotherapy, HIPEC, anti-PD-1 and anti-HER-2 therapy, which will provide a clinical basis for the treatment of advanced GC.

DETAILED DESCRIPTION:
Gastric cancer (GC) is the 5th most common malignant tumor worldwide, and it causes the 4th most tumor-related deaths among all malignant tumors. China is a large country with 40% of the total number of GC cases worldwide. Despite the advances in medical detection methods, most of the GC patients in China are in the advanced stage at the time of diagnosis, in which peritoneal metastasis is one of the common metastatic patterns of advanced GC, and the presence of peritoneal metastasis accounts for about 46% of patients with distant metastasis detected at the first diagnosis. The prognosis of GC patients with peritoneal metastasis is extremely poor, and compared with other metastatic organs, patients with stage IV GC with peritoneal metastasis have a worse prognosis and shorter survival.

The treatment of peritoneal metastasis of GC has been based on systemic chemotherapy with reference to advanced GC, but it is difficult for traditional chemotherapeutic agents to reach the peritoneal lesions due to the existence of blood-peritoneal barrier. In recent years, heat intraperitoneal perfusion chemotherapy (HIPEC) has gained better efficacy in the treatment of peritoneal metastases of many malignant tumors, including GC.HIPEC allows chemotherapeutic drugs to act directly on tumor tissues while reducing the impact on other parts of the body; the warming effect is synergistic with the antitumor effects of chemotherapeutic drugs and helps the drugs to act more efficiently on the intraperitoneal tumor cells; moreover, the chemotherapeutic drugs are absorbed through the peritoneum and then enter the liver via the portal vein route, which is beneficial to preventing liver metastasis. HIPEC currently has four applications and indications in the clinic: firstly, palliative application to improve the quality of life for GC abdominal metastasis with a large amount of carcinomatous ascites; secondly, therapeutic application of radical gastric cancer surgery + cytoreductive surgery + HIPEC for the treatment of GC; third, prophylactic application, radical gastric cancer surgery + peritoneal hyperthermia chemotherapy, targeting people with high risk of peritoneal recurrence, especially patients with T3-4 or positive lymph nodes; fourth, neoadjuvant application, neoadjuvant chemotherapy combined with peritoneal hyperthermia chemotherapy before radical gastric cancer treatment, in order to reduce the risk of peritoneal implantation of gastric cancer and to increase the possibility of radical surgery. However, there is a lack of high-level evidence-based medical evidence on the efficacy and safety of HIPEC as a translational treatment for GC with peritoneal metastasis.

The use of immune checkpoint inhibitors (ICIs) in the treatment of advanced GC has made significant progress in recent years. The KEYNOTE series of studies evaluated the safety and efficacy of PD-L1 antibody as a first-line treatment for advanced GC, among which the results of KEYNOTE-859 confirmed that the combination of Pembrolizumab and chemotherapy is expected to be a HER-2 negative advanced gastric/esophagogastric junctional cancer first-line treatment option. A recent retrospective study by Chinese scholars demonstrated that patients with stage IV GC who were responded to the immunotherapy combined with chemotherapy as the first-line treatment were able to achieve significant survival benefit after radical resection. However, whether HIPEC combined with immunotherapy for peritoneal metastatic gastric cancer improves the R0 resection rate and prolongs survival time is currently unclear.

Therefore, we conducted this prospective multicenter clinical trial trying to combine the specificity of HIPEC for peritoneal metastases with immunotherapy for advanced GC, aiming to evaluate the efficacy and feasibility of multimodal treatment regimens, such as HIPEC in combination with immunotherapy, for the transformative treatment of peritoneal metastases of GC or EJ junctional cancer and to explore the effective dose and safety of the combination of systemic chemotherapy, HIPEC, anti-PD-1 and anti-HER-2 therapy, which will provide a clinical basis for the treatment of advanced GC.

ELIGIBILITY:
Inclusion Criteria:

1. patients with a pathologically confirmed primary diagnosis of gastric/esophagogastric junctional cancer who have not undergone chemotherapy, radiotherapy, or other antitumor therapy prior to the start of the clinical trial;
2. age 18 to 75 years Eastern Coorperative Oncology Group (ECOG): 0 to 1 points;
3. diagnosis of metastatic adenocarcinoma of the peritoneum [peritoneal cancer index (PCI) ≤ 20 points] with or without ascites (beyond the pelvis but not reaching full abdominal ascites) by laparoscopic exploration;
4. Voluntarily sign the informed consent form.
5. good cardiac function for resection with curative intent. If clinically indicated, patients with underlying ischemic, valvular heart disease or other severe heart disease should be evaluated preoperatively by a cardiologist;
6. normal function of major organs and subjects are required to meet the following laboratory criteria: 1) Absolute neutrophil count (ANC) ≥ 1.5x109/L in the last 14 days without granulocyte colony-stimulating factor (GCSF); 2) Platelets ≥ 100 x 109/L in the absence of blood transfusion in the last 14 days; 3) Hemoglobin > 9 g/dL without transfusion or erythropoietin use in the last 14 days; 4) Total bilirubin ≤ 1.5 x upper limit of normal (ULN); enrollment is also allowed if total bilirubin > 1.5 x ULN but direct bilirubin ≤ ULN; 5) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN.

6) Blood creatinine ≤1.5×ULN and creatinine clearance (calculated using the Cockcroft-Gault formula) ≥60 ml/min; 7) good coagulation function, defined as International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 x ULN; 8) Normal thyroid function, defined as thyrotropin (TSH) within the normal range. If baseline TSH is outside the normal range, subjects may also be enrolled if total T3 (or FT3) and FT4 are within the normal range; 9) Cardiac enzyme profiles within the normal range (enrollment will be allowed if the investigator determines that the laboratory abnormality is not of clinical significance); 7) Thyroid function: thyroid stimulating hormone (TSH) and free thyroxine (FT3/FT4) in the normal range or mildly abnormal without clinical significance; 8. weight of 40 kg or more (including 40 kg), or BMI > 18.5; 9. female patients must meet:

* Menopausal (defined as absence of menstruation for at least 1 year with no confirmed cause other than menopause) status, or surgically sterilized (removal of ovaries and/or uterus), or patients of childbearing potential must also meet the following requirements:
* Pregnancy test within 7 days prior to first dose must be negative;
* Agree to use contraception with an annual failure rate of < 1% or remain abstinent (avoid heterosexual intercourse) (at least 120 days from signing the informed consent form until at least 9 months after the last dose of the test drug and at least 9 months after the procedure (contraceptive methods with an annual failure rate of < 1% include bilateral tubal ligation, male sterilization, proper use of hormonal contraceptives that suppress ovulation, hormone-releasing intrauterine contraceptives, and copper-containing intrauterine devices). .;
* No breastfeeding is allowed. 10. The subject reads and fully understands the patient instructions and signs the informed consent form.

Exclusion Criteria:

1. the patient has a previous (within 5 years) or concurrent other malignant tumor;
2. patients who are preparing for or have previously received organ or bone marrow transplantation;
3. have had a blood transfusion within 2 weeks prior to the first dose, or have a history of bleeding, and any bleeding event with a severity rating of 3 or more on the CTCAE 4.0 within 4 weeks prior to screening;
4. abnormal coagulation with bleeding tendency (INR in the absence of anticoagulants at normal values > 1.5); patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin, or their analogues; the use of low-dose warfarin (1 mg orally once daily) for prophylactic purposes is permitted, provided the International Normalized Ratio of the prothrombinogen time (INR) is ≤ 1.5, or Small-dose aspirin (no more than 100 mg daily);
5. an actinic/venous thrombotic event within 6 months prior to screening, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis (except for venous thrombosis due to intravenous cannulation for pre-chemotherapy, which has resolved in the judgment of the investigator), and pulmonary embolism;
6. myocardial infarction, poorly controlled arrhythmia (including QTc interval ≥ 450 ms in men and ≥ 470 ms in women) within 6 months prior to the first dose (QTc interval is calculated using the Fridericia formula);
7. the presence of NYHA class III-IV cardiac insufficiency or cardiac ultrasound: LVEF (left ventricular ejection fraction) <50%;
8. urine protein ≥++ and confirmed 24-hour urine protein quantification >1.0 g;
9. have multiple factors that interfere with oral administration of medications (e.g., inability to swallow, chronic diarrhea, and intestinal obstruction)
10. pleural effusion with clinical symptoms requiring clinical intervention;
11. human immunodeficiency virus (HIV) infection;
12. active tuberculosis;
13. long-standing unhealed wounds or incompletely healed fractures;
14. patients with pre-existing and current interstitial pneumonitis, pneumoconiosis, radiation pneumonitis, drug-associated pneumonitis, and severely impaired lung function that may interfere with the detection and management of suspected drug-associated pulmonary toxicity
15. the presence of a known active or suspected autoimmune disease, except those who are in a stable state of that disease at the time of enrollment (not requiring systemic immunosuppressive therapy);
16. a history of severe chronic autoimmune disease, such as systemic lupus erythematosus; a history of inflammatory bowel disease, such as ulcerative enteritis, Crohn's disease, or chronic diarrheal disease, such as irritable bowel syndrome; a history of tuberculosis or tuberculosis; a history of active hepatitis B, hepatitis C, or HIV; or well-controlled non-severe immune disorders, such as dermatitis, arthritis, or psoriasis, may be eligible. .. Hepatitis B virus titers < 500copy/ml may be enrolled;
17. patients requiring treatment with systemic corticosteroids (> 10 mg/day prednisone efficacy dose) or other immunosuppressive drugs within 14 days prior to the first dose or during the study period. However, enrollment is permitted if patients are allowed to use topical topical or inhaled steroids, or adrenal hormone replacement therapy at doses ≤ 10 mg/day prednisone efficacy dose in the absence of active autoimmune disease;
18. any active infection requiring systemic administration of anti-infective therapy within 14 days prior to the first dose; except for prophylactic antibiotic therapy (e.g., for the prevention of urinary tract infections or chronic obstructive pulmonary disease);
19. treatment with a live vaccine within 28 days prior to the first dose; except inactivated viral vaccines for seasonal influenza;
20. prior treatment with antibodies/drugs targeting immune checkpoints, e.g., PD-1, PD-L1, CTLA-4 inhibitors, etc;
21. have received treatment with immunologically-affecting related drugs or medical technologies (including but not limited to the following: thymopentin, thymofacine, interferon, CAR-T therapy, etc.) within 6 months prior to the first dose of the drug
22. is receiving treatment in another clinical study or is scheduled to begin treatment in this study less than 1 month from the end of treatment in the previous clinical study;
23. has a known history of allergy or intolerance to any study medication or its components
24. patients with a history of alcoholism, drug abuse, and substance abuse. Patients who have stopped drinking alcohol may be enrolled;
25. patients with non-compliance with medical advice, non-adherence to prescribed medication, or incomplete information that may affect the judgment of efficacy or safety;
26. pregnant or lactating female patients;
27. patients with conditions that may increase the risk of study participation and study medication, or other severe, acute, and chronic conditions that, in the judgment of the investigator, make participation in a clinical study unsuitable.
28. other conditions that, in the judgment of the investigator, make them unsuitable for this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 1 year
  The proportion of patients still alive at one year from the start of patient enrollment was calculated as a percentage of all patients. Deaths from all causes were included in the calculation of overall survival. The OS of patients who did not reach the one-year loss to follow-up was counted as data censored at the time of last confirmed survival before the loss to follow-up, i.e., only the time point of last known survival was counted in the number of survivors.

SECONDARY OUTCOMES:
Progression-free Survival | 1 year
  Percentage of all patients who did not experience disease progression or death within one year from the start of patient enrollment. If disease progression is indicated by imaging, the date of disease progression will be the time of the imaging exam that clearly confirms disease progression. If disease progression was diagnosed by other clinical modalities, the date of diagnosis will be used as the date of disease progression. Patients who discontinued the trial (without follow-up imaging) for reasons other than disease progression and patients who received post-trial therapy will have the time of discontinuation of the trial or the time of initiation of post-trial therapy as the data censored. New onset of other tumors is not considered a disease progression event and is also not censored as data.
Completeness of cytoreduction score | 1 year
  CC-0 indicates no residual tumor visible to the naked eye, CC-1 indicates residual tumor with a maximum diameter of <2.5 mm, CC-2 indicates residual tumor with a diameter of more than 2.5 mm but <25 mm, and CC-3 indicates residual tumor with a diameter of ≥25 mm. CC-0 and CC-1 are usually classified as complete cytoreduction.
Objective Response Rate | 1 year
  Refers to the proportion of patients whose tumors shrank to a certain level and remained there for a certain period of time, and includes both CR (Complete Response) and PR (Partial Response) cases. Objective tumor remission was assessed using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). Patients had to be accompanied by measurable tumor lesions at baseline, and the efficacy assessment criteria were classified as Complete Response (CR), Partial Response (PR), Stable Disease (SD), and Progressed Disease (PD) according to the RECIST 1.1 criteria. Disease (PD).

CONTACTS AND LOCATIONS:
Overall Officials: Zekuan Xu, PhD, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
The data and materials of the study will be made available on request.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Zhang Y, Li F, Liu H, Li P, Li Q, Wang L, Zhang D, Wu H, Xu H, Yang L, Xu ZK. Efficacy and safety of HIPEC combined with PD-1 and SOX chemotherapy for gastric or oesophagogastric junctional cancer with peritoneal metastasis (HISTORIA): protocol for a prospective, multicentre, single-arm, phase II study. BMJ Open. 2025 Sep 14;15(9):e098326. doi: 10.1136/bmjopen-2024-098326. PMID 40953882